CLINICAL TRIAL: NCT05199753
Title: A Phase I/II, First-in-Human (FIH), Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LM-108 as a Single Agent or in Combination With Anti-PD-1 Antibody in Subjects With Advanced Solid Tumours
Brief Title: Study of LM-108 as a Single Agent or in Combination With Anti-PD-1 Antibody in Subjects With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Australia Pty Limited (Industry)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM108-01-101
Record Dates: First submitted 2021-12-15; First posted 2022-01-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LM-108 Dose Escalation (Experimental)
  Interventions: Drug: LM-108
- LM-108 Dose Expansion (Experimental)
  Interventions: Drug: LM-108
- LM-108 combination dose escalation (Experimental)
  Interventions: Drug: LM-108; Drug: An Anti-PD-1 Antibody
- LM-108 combination dose expansion (Experimental)
  Interventions: Drug: LM-108; Drug: An Anti-PD-1 Antibody

INTERVENTIONS:
Drug: LM-108 — Administered intravenously
Drug: An Anti-PD-1 Antibody — Administered intravenously
  Arms: LM-108 combination dose escalation; LM-108 combination dose expansion

SUMMARY:
This is a first-in-human, Phase I/II, open-label, multi-centre, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumour activity of LM-108 as a single agent or in combination with an anti-PD-1 mAb in subjects with solid tumours.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
2. Histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
3. At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
4. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose

Key Exclusion Criteria:

1. Any adverse event from prior anti-tumour therapy has not yet recovered to ≤grade 1 of CTCAE v5.0
2. Uncontrolled tumour-related pain
3. Known central nervous system (CNS)
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
5. Use of inhaled corticosteroids
6. Known history of autoimmune disease
7. Use of any live attenuated vaccines within 28 days
8. Have severe cardiovascular disease
9. Uncontrolled or severe illness
10. History of immunodeficiency disease
11. Active malignancies which are likely to require the treatment.
12. Child-bearing potential female
13. Have psychiatric illness or disorders

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 126 weeks
Incidence of dose-limiting toxicity (DLT) | 126 weeks
Incidence of serious adverse event (SAE) | 126 weeks
Incidence of clinical significant in laboratory examinations, including hematology, urinalysis, blood biochemistry, coagulation tests and thyroid function. | 126 weeks

SECONDARY OUTCOMES:
Incidence of anti-drug antibodies to LM-108 | 126 weeks
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) for LM-108 | 126 weeks
PK Parameter: Minimum Observed Concentration (Cmin) for LM-108 | 126 weeks
PK Parameter: Time of Maximum Observed Concentration (Tmax) for LM-108 | 126 weeks
PK Parameter: Area Under the Concentration-time Curve (AUC) for LM-108 | 126 weeks
PK Parameter: Steady State Maximum Concentration (Cmax,ss) | 126 weeks
PK Parameter: Steady State Minimum Concentration (Cmin, ss) | 126 weeks
PK Parameter: Systemic Clearance at Steady State (CLss) | 126 weeks
PK Parameter: Accumulation Ratio (Rac) | 126 weeks
PK Parameter: Elimination Half-life (t 1/2) | 126 weeks
PK Parameter: Volume of Distribution at Steady-State (Vss) | 126 weeks
PK Parameter: Degree of Fluctuation (DF) | 126 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Blacktown Hospital, Sydney, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - ICON Cancer Centre, South Brisbane, Queensland
  - Cabrini Health Limited, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - One Clinical Research Pty Ltd., Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No